CLINICAL TRIAL: NCT05838898
Title: Changes of Corneal Endothelial Cells in Patients With PDR Using Specular Microscopy
Brief Title: Specular Microscopy in Patients With Proliferative Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marline Reda Fahim Anis, Ophthalmologist, Assiut University
Other Study IDs: Specular microscopy
Record Dates: First submitted 2022-09-09; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Corneal Endothelial Cell Changes in Diabetic Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Specular microscopy — Non-contact Specular microscopy is a non-invasive method that allows for in vivo study of corneal endothelium.

SUMMARY:
.1. corneal endothelial profile in patients with proliferative diabetic retinopathy compared to a healthy age-matched control group.

2. The effect of the age, and duration of Diabetes on the corneal endothelium .

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a group of metabolic diseases characterized by hyperglycemia resulting from defects in insulin secretion, insulin action, or both. The chronic hyperglycemia of diabetes is associated with long-term damage, dysfunction, and failure of different organs, especially the eyes, kidneys, nerves, heart, and blood vessels. In Egypt, diabetes is a growing public health problem.

Diabetes causes several ocular complications including diabetic retinopathy, cataract, glaucoma and ocular surface diseases.

Retinal damage caused by microangiopathy results in diabetic retinopathy which is one of the most important causes of blindness and affects approximately 40% of all diabetic patients.

Diabetic retinopathy is classified to non-proliferative diabetic retinopathy (NPDR) (mild, moderate, severe) and proliferative diabetic retinopathy (PDR) according to the severity of retinopathy.

Even though diabetic retinopathy is the most common sequel and most widely studied association of DM, other structures of the eye are not immune and get affected in various stages of the disease.

Chronic hyperglycemia can affect the corneal layers shape and functions. The resultant morphological and functional alterations increase the susceptibility of the cornea to recurrent corneal erosions, superficial keratitis, punctate epithelial keratopathy, impaired corneal sensitivity, and slowed healing capacity following trauma or surgical insult.

Considering the pivotal role of corneal endothelium in maintaining corneal clarity, several studies have investigated the possible alterations that take place in corneal endothelium in patients with DM . These studies found that DM can cause structural changes in corneal endothelial cells . Damaged corneal endothelium results in corneal oedema and increased central corneal thickness (CCT) . This increase has been documented in patients with DM as compared with healthy controls in a number of studies .

The aim of this study is to investigate the corneal endothelial cell profile and central corneal thickness in patients with proliferative diabetic retinopathy using non-contact specular microscopy.

ELIGIBILITY:
Inclusion Criteria:

* patients with Type I or II Diabetes Mellitus

.Diagnosed with proliferative diabetic retinopathy . .Intraocular pressure less than 21mmHg.

Healthy controls:

.Healthy individuals aged 40 to 70 years of both sexes. .Intraocular pressure less than 21 mmHg.

Exclusion Criteria:

* Diabetic group:
* Associated ocular diseases that may affect the corneal endothelium such as uveitis, glaucoma, and dystrophy, prolonged CLs use.
* Previous ocular trauma or surgery.

Healthy control:

* Any systemic diseases that may affect corneal endothelium function.
* Associated ocular diseases that may affect the corneal endothelium such as uveitis, glaucoma, and dystrophy, prolonged CLs use.
* Previous ocular trauma , surgery ,laser or intraocular injection.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Image capture will be done by the same individual for all subjects. The following data will be collected and analyzed: corneal endothelial cell count, coefficient of variation, percentage of hexagonal cells and central corneal thickness.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To predict the effect of Diabetes on the cornea of diabetic patients | Baseline
  To evaluate corneal endothelial changes in patients with Proliferative diabetic retinopathy compared to normal group of the same age and gender using Specular microscopy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mortazavi SA, Akhlaghi M, Dehghani A, Pourazizi M, Malekahmadi M, Fazel M, Tavakoli M, Noorshargh P. Diabetic retinopathy and corneal endothelial parameters: an analytical cross-sectional study. BMC Ophthalmol. 2022 Nov 9;22(1):427. doi: 10.1186/s12886-022-02667-6. PMID 36348282
- [Background] Jha A, Verma A, Alagorie AR. Association of severity of diabetic retinopathy with corneal endothelial and thickness changes in patients with diabetes mellitus. Eye (Lond). 2022 Jun;36(6):1202-1208. doi: 10.1038/s41433-021-01606-x. Epub 2021 Jun 11. PMID 34117392